CLINICAL TRIAL: NCT01999088
Title: Randomized, Double-blind, Cross-over Placebo-controlled Study to Assess the Functional Meat Products With n-3 and Rosemary Extract Fluid in Biochemical Markers of Cardiovascular Disease Related Risk in Subjects at Low Risk for Cardiovascular Disease
Brief Title: Health Benefits of Functional Meat (With n-3 Fatty Acids and Rosemary Extract) on Low Risk for Cardiovascular Disease People
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Spanish Ministry of industry, tourism and trade (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: HULP-2889
Record Dates: First submitted 2013-11-19; First posted 2013-12-03 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-11

CONDITIONS: Low Risk for Cardiovascular Disease
Keywords: Fatty Acids, Omega-3; Rosemary extract; Functional meat; Cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Functional Food; Hazard Analysis and Critical Control Points

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Functional meat (Experimental): During the I period, volunteers weekly consumed three 150g/serving Functional Meat (FM) products (cooked Ham and Turkey breast). It was firmly recommended that all other meats and meat derivatives had to be excluded from the diet.
  Interventions: Other: Functional Meet; Other: Control Meat
- Control Meat (Placebo Comparator): During the C period, volunteers consumed identical amounts of meat products that did not include functional ingredients (Control Meat (CM)).
  Interventions: Other: Functional Meet; Other: Control Meat

INTERVENTIONS:
Other: Functional Meet — During the I period, volunteers weekly consumed three 150g/serving Functional Meat (FM) products (cooked Ham and Turkey breast). It was firmly recommended that all other meats and meat derivatives had to be excluded from the diet.
  Other Names: Functional food
Other: Control Meat — During the C period, volunteers consumed identical amounts of meat products that did not include functional ingredients (Control Meat (CM)).
  Other Names: Control Food

SUMMARY:
Volunteers were randomly assigned by gender to follow of two 12 weeks experimental periods: intervention (I) and control (C) in different order (I/C or C/I). Both periods were separated by a 4 weeks wash-out interval during which subjects returned to their usual diet:

During the I period, volunteers weekly consumed three 150g/serving Functional Meat (FM) products (cooked Ham and Turkey breast). It was firmly recommended that all other meats and meat derivatives had to be excluded from the diet.

During the C period, volunteers consumed identical amounts of meat products that did not include functional ingredients (Control Meat (CM)).

Functional meat (FM) products (Functional cooked Ham (FH) and Functional cooked Turkey breast (FT)), were manufactured mixing the meats with the patented formula® (P200402755.2004). The amount of supercritical rosemary extract, deodorized salmon oil and vitamin E used was respectively, 0.02% w/w, 0.6% w/w, and 0.001% w/w.

Control meat (CM) products (Control cooked Ham (CH) and Control cooked Turkey (CT), were prepared without addition of the functional ingredients.

DETAILED DESCRIPTION:
The total duration of the study was 28 weeks: first experimental period 0-12 weeks, washout period 12-16 weeks second experimental period 16-28 weeks:

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged over 18 years
* At least 2 lipid profile parameters altered (TAG ≥150 mg /dl and/or total cholesterol ≥200 mg / dl and/or LDL ≥130 mg / dl and/or HDL ≥40mg/dl men or ≥ 50mg/dl women).
* Signed informed consent

Exclusion Criteria:

* Individuals with body mass index (BMI) ≥ 35 kg/m2
* Individuals with Diabetes Mellitus insulin dependent
* Individuals with disorders associated with eating behaviour
* Individuals with consumption of omega 3 functional foods, fish oil or antioxidant supplements
* Individuals inability to consume the test foods (ej. Vegetarians)
* Individuals with special diet due to disease as celiac disease, chronic renal failure, etc.
* Individuals with mental disease or low cognitive function.
* Individuals with consumption of drugs to weight lost.
* Individuals treated with drugs whose direct effect is on lipid profile (statins, fibrates, diuretics, corticosteroids or oral anti-inflammatory).
* Individuals with diseases that could be involucrate in weight lost (not controlled hypothyroidism, serious psychiatric illness, etc.).
* Pregnant women or lactating.
* Individuals with regular consumption of anti-inflammatory or glucocorticoids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Lipid profile changes | 0, 12, 16 and 28 week
  Parameters measured were: Cholesterol, LDL-Cholesterol, HDL-Cholesterol, Triglycerides, Apolipoprotein B and Apolipoprotein A.

SECONDARY OUTCOMES:
Framingham score changes | 0, 12, 16 and 28 week
  Framingham score adapted to Spanish population (cardiovascular risk measurement)
Inflammatory markers changes | 0, 12, 16 and 28 week
  Parameters measured were: Adiponectin, fibrinogen, TNFα, IL6, IL1B, PAI-1 and PCR
Oxidative Stress Parameters changes | 0, 12, 16 and 28 week
  Parameters measured were: plasma antioxidant capacity (FRAP, ferric reducing antioxidant power), lipidic peroxidation (TBARS, thiobarbituric acid reactive substances assay), LDL-ox, . 8-iso-Prostaglandin F2α (8-iso-PGF2α), α-tocopherol and nitric oxide synthase (NOS).
Glucosa Metabolism changes | 0, 12, 16 and 28 week
  Parameters measured were: glucose, basal insulin, HOMA index (glycemic insulin sensitivity index was calculated using the formula: HOMA-IR = fasting glucose (mmol/l)/fasting immunoreactive insulin (mU/ml)/22.5).
Blood pressure and heart rate changes | 0, 12, 16 and 28 week
Anthropometric parameters changes | 0, 12, 16 and 28 week
  Parameters measured were: Weight, Height and waist circumference, tricipital skinfold thickness and fat mass percentage (FM%).

OTHER OUTCOMES:
Homocystein levels changes | 0, 12, 16 and 28 week
Sensory perception | 12, and 28 week
  Subjects were asked to value taste and smell meats consumed, using a Visual Analogical Scale ranged 1-10 cm.
Adverse event | 12, and 28 week
  Defined as any unfavourable, unintended effect reported by a subject or observed by the investigator during the study. All were recorded along with the symptoms involved (nausea, vomiting, diarrhoea, halitosis, constipation).

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Gomez-Candela, MD, PhD, Principal Investigator — Hospital Universitario La Paz
Locations (1):
- Hospital Universitario La Paz, Madrid, Maadrid, Spain

REFERENCES:
- [Derived] Bermejo LM, Lopez-Plaza B, Weber TK, Palma-Milla S, Iglesias C, Reglero G, Gomez-Candela C. Impact of cooked functional meat enriched with omega-3 fatty acids and rosemary extract on inflammatory and oxidative status; a randomised, double-blind, crossover study. Nutr Hosp. 2014 Nov 1;30(5):1084-91. doi: 10.3305/nh.2014.30.5.8048. PMID 25365012
- See also: Institute for Health Research IdiPAZ — http://www.idipaz.es